CLINICAL TRIAL: NCT04353375
Title: An Open-Label, Single-Arm, Multicenter Phase 2/3b Clinical Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of HMPL-453 Tartrate in Patients With Advanced Intrahepatic Cholangiocarcinoma Habouring FGFR2 Fusion/Rearrangement
Brief Title: HMPL-453 Tartrate in Advanced Intrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-453-00CH2
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Advanced Intrahepatic Cholangiocarcinoma; Solid Tumor, Adult
Keywords: FGFR2 funsion; HMPL-453; ICC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HMPL-453 (Experimental): HMPL-453 150mg QD HMPL-453 300mg QD
  Interventions: Drug: HMPL-453

INTERVENTIONS:
Drug: HMPL-453 — Cohort_1:HMPL-453 150mg QD continuously in 21-day cycles; Cohort_2, Cohort_3 and Cohort_4:HMPL-453 tartrate 300 mg QD orally (for 14 consecutive days [Day 1 to 14], followed by 7 days off [Day 15 to 21], 21 days as a treatment cycle)

SUMMARY:
The goal of this clinical trial is to evaluate in patients with advanced intrahepatic cholangiocarcinoma harboring FGFR2 fusion/rearrangement. The main questions it aims to answer are:

To evaluate the objective response rate (ORR) of HMPL-453 tartrate in the treatment of patients with advanced intrahepatic cholangiocarcinoma (ICC) habouring fibroblast growth factor receptor (FGFR) 2 fusions/rearrangements after at least one line of systemic treatment failure or intolerance Participants will receive HMPL-453 tartrate 300 mg QD orally (for 14 consecutive days [Days 1 to 14] followed by 7 days off [Day 15 to 21], 21 days as a treatment cycle.]

DETAILED DESCRIPTION:
This is an open-label, single-arm, multicenter phase 2/3b clinical study to evaluate the efficacy and safety of HMPL-453 tartrate in the treatment of patients with advanced ICC habouring FGFR2 fusions/rearrangements/mutations. The study consists of the following 4 cohorts.

Cohort 1: Approximately 12 patients with locally advanced unresectable or metastatic ICC habouring FGFR2 fusions/rearrangements after at least one line of systemic treatment failure or intolerance are planned to be enrolled in this cohort to receive HMPL-453 tartrate 150 mg administered orally once daily (QD) continuously in 21-day cycles.

Cohort 2: A total of approximately 113-116 patients are planned to be enrolled in this cohort, divided into safety run-in and extension phases. Approximately 6 to 9 patients with solid tumors who failed standard treatment or had intolerable toxicity will be enrolled into the first phase (safety run-in phase), to receive HMPL-453 tartrate 300 mg QD orally (for 14 consecutive days [Day 1 to 14], followed by 7 days off [Day 15 to 21], 21 days as a treatment cycle). Dose limiting toxicities (DLT) observation period consists of 28 days, in which a cycle of treatment will be received. Patients will enter second stage of cohort 2 (extension phase) after completion of safety run-in assessments. Approximately 20 patients with locally advanced unresectable or metastatic ICC habouring FGFR2 fusions/rearrangements after at least one line of systemic treatment failure or intolerance will receive HMPL-453 tartrate 300 mg QD orally administered (for 14 consecutive days [Day 1 to 14], followed by 7 days off [Day 15 to 21], 21 days as a treatment cycle). Based on the efficacy and safety data of the enrolled patients, and after reaching an agreement with China Center for Drug Evaluation on 17 Feb 2023, approximately 87 patients with locally advanced unresectable or metastatic ICC habouring FGFR2 fusions/rearrangements after at least one line of systemic treatment failure or intolerance will be enrolled to support registration submission as the registration study stage of this study, receiving HMPL-453 tartrate 300 mg QD orally (for 14 consecutive days [Days 1 to 14] followed by 7 days off [Day 15 to 21], 21 days as a treatment cycle.

Cohort 3 (Confirmatory Study Cohort): A total of approximately 87 patients with locally advanced unresectable or metastatic ICC harbouring FGFR2 fusions/rearrangements after at least one line of systemic treatment failure or intolerance are planned to be enrolled in this cohort, as the confirmatory study phase of this study. Patients will receive HMPL-453 tartrate 300 mg QD for 14 days (Days 1 to 14), followed by 7 days off (Days 15 to 21), (21-day treatment cycles).

Cohort 4 (Exploratory Cohort): Approximately 10 to 20 treatment-naïve patients with locally advanced unresectable or metastatic ICC harbouring FGFR2 fusions/rearrangements/mutations are planned to be enrolled in this cohort. Patients will receive HMPL-453 tartrate 300 mg QD orally for 14 days (Days 1 to 14), followed by 7 days off (Days 15 to 21) (21-day treatment cycles).

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood the study and voluntarily signed the ICF;
2. Age ≥ 18 years;
3. a. pathologically or cytologically confirmed advanced treatment failure solid tumor with standard patients (applicable to cohorts2 stage I); b. histologically or cytologically confirmed histologically or cytologically confirmed locally advanced unresectable or metastatic ICC patients with FGFR2 fusions/rearrangements/mutation (applicable to Cohort 1, Cohort 2 Stage II, Cohort 3 and Cohort 4)
4. a. The patients have received at least one prior systemic treatment regimen for advanced ICC and has intolerable PD or toxicity(Cohort1-3); b. Patients who have not received any prior systemic therapy for advanced ICC(Cohort4)
5. Measurable lesion according to RECIST v1.1;
6. ECOG performance status of 0 or 1;
7. Life expectancy ≥ 12 weeks;
8. Female patients or male patients with partners of childbearing potential must take effective contraceptive measures per the protocol.

Exclusion Criteria:

1. Patients who previously received selective FGFR targeting therapy;
2. Received approved or researched systemic anti-tumor treatment within 3 weeks prior to the start of the study treatment;
3. Radical radiotherapy within 4 weeks;
4. Have received local anti-tumor treatment within 4 weeks;
5. Major surgery requiring hospitalization or incomplete healing of the surgery incision within 4 weeks;
6. Current or prior history of retinal detachment;
7. Using a strong inducer or inhibitor of cytochrome P450 3A (CYP3A) within 2 weeks or 5 half-lives of the study treatment;
8. Taking drugs or dietary supplementsthat may cause blood phosphorus and/or blood calcium to rise within 2 weeks prior to the start of the study treatment;
9. International normalized ratio above 1.5 or partial activated prothrombin time above 1.5 times ULN;
10. History of clinically significant active hepatopathy, including active viral hepatitis, or other active hepatitis, clinically significant moderate to severe liver cirrhosis;
11. The patients with human immunodeficiency virus (HIV) infection;
12. Active infection requiring systemic treatment within 1 week prior to the start of the study treatment;
13. Screening blood phosphorus levels above ULN, or history of abnormal calcium phosphorus metabolism requiring clinical intervention or relevant medical history;
14. Currently keratopathy confirmed by ophthalmological examination;
15. Prior history of retinal detachment, or current diseases that may cause retinal detachment;
16. Clinically significant arrhythmia or conduction abnormalities requiring clinical intervention;
17. Patients with known deep venous thrombosis, treated with low molecular weight heparin (LMWH) or drugs with similar efficacy, and the investigator judges that the thrombosis is stable for ≥ 2 weeks ;
18. Toxicities caused by prior anti-tumor treatment have not recovered to grade 0 or 1;
19. The patient has any current disease or condition that affects drug absorption, or the patient cannot be orally administered;
20. Combined with other malignant tumor or a history of other malignant tumor within 5 years prior to study screening;
21. Patients currently has central nervous system metastases, meningeal metastases or spinal cord compression, except in individual cases;
22. Any other medical condition or clinically significant laboratory abnormalities judged by the investigator would make the patients unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Measured up to 6 months after the last patient has been enrolled or all patients have finished their last PFS follow up, whichever comes first
  Proportion of patients whose best overall response are confirmed CR or PR

SECONDARY OUTCOMES:
Disease control rate (DCR) | Measured up to 6 months after the last patient has been enrolled or all patients have finished their last PFS follow up, whichever comes first
  Proportion of patients whose best overall response after treatment is confirmed CR or PR, or judged as SD (SD≥6 weeks)
Time to response (TTR) | Measured up to 6 months after the last patient has been enrolled or all patients have finished their last PFS follow up, whichever comes first
  The time from the first dose of study drug to the first CR or PR in patients whose best overall response is a confirmed CR or PR
Duration of response (DoR) | Measured up to 6 months after the last patient has been enrolled or all patients have finished their last PFS follow up, whichever comes first
  The time from initial CR or PR to PD or death from any cause, whichever comes first, in patients whose best overall response is a confirmed CR or PR
Progression-Free Survival (PFS) | Measured up to 6 months after the last patient has been enrolled or all patients have finished their last PFS follow up, whichever comes first
  The time from the first study treatment to the onset of PD or death from any cause
Overall survival (OS) | up to 2 years
  The time from the patients receiving the first study drug until the death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, PhD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No